CLINICAL TRIAL: NCT02455102
Title: Electronic Warning System to Improve Stroke Prevention in Atrial Fibrillation - A Quality Improvement Initiative at the University Hospital Bern
Brief Title: Electronic Warning System for Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 022/14
Record Dates: First submitted 2015-05-06; First posted 2015-05-27 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Atrial Fibrillation
Keywords: Prevention; Anticoagulation; Electronic warning system
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electronic alert (Active Comparator): Physicians, whose patients with atrial fibrillation do not receive stroke preventive measures, will receive an electronic warning alert.
  Interventions: Other: Electronic warning alert
- No electronic alert (No Intervention): Physicians, whose patients with atrial fibrillation do not receive stroke preventive measures, will receive no electronic warning alert.

INTERVENTIONS:
Other: Electronic warning alert — A newly-installed warning system for stroke prevention in atrial fibrillation.
  Arms: Electronic alert

SUMMARY:
The aim of this randomized controlled study is to evaluate whether a newly designed electronic warning system will increase the initiation rate of adequate stroke preventive measures in patients with atrial fibrillation.

DETAILED DESCRIPTION:
A large proportion of patients with atrial fibrillation do not receive stroke prevention therapy in line with the guidelines, in spite of the presence of an increased risk of stroke. It will be investigated whether an electronic alert to physicians, whose patients with atrial fibrillation do not receive stroke preventive measures, will increase the rate of adequate stroke preventive measures as compared to a control group of patients without an electronic alert. The electronic alerts will be sent if patients with atrial fibrillation but without adequate stroke preventive measures receive in-patient treatment at the University Hospital Bern. The electronic alert system includes a feature that helps the physicians in charge to evaluate the CHA2DS2VASC Score. At the end of the hospital stay medical discharge letters will be reviewed for initiation of adequate stroke preventive measures.

ELIGIBILITY:
Inclusion Criteria:

* All in-patients with atrial fibrillation

Exclusion Criteria:

* Ongoing anticoagulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1707 (Actual)
Dates: Start 2014-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Rate of initiation of adequate measures to prevent stroke (oral anticoagulant prescription) by physician in charge | End of hospital stay (expected average duration of 1 week)
  Reviewed from discharge letter

SECONDARY OUTCOMES:
Use of the CHA2DS2VASc score calculation tool by the physician in charge | During hospital stay (expected average duration of 1 week)
Rate of correct evaluation of the CHA2DS2VASC Score through the calculation tool by physician in charge | End of hospital stay (expected average duration of 1 week)

CONTACTS AND LOCATIONS:
Overall Officials: Nils Kucher, Prof. M.D., Principal Investigator — Department of Angiology, Swiss Cardiovascular Center, University of Berne
Locations (1):
- Swiss Cardiovascular Center, Inselspital, University of Bern, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Derived] Silbernagel G, Spirk D, Hager A, Baumgartner I, Kucher N. Electronic Alert System for Improving Stroke Prevention Among Hospitalized Oral-Anticoagulation-Naive Patients With Atrial Fibrillation: A Randomized Trial. J Am Heart Assoc. 2016 Jul 22;5(7):e003776. doi: 10.1161/JAHA.116.003776. PMID 27451467